CLINICAL TRIAL: NCT03928145
Title: Efficacy of Chlorthalidone and Hydrochlorothiazide in Combination With Amiloride in Multiple Doses on Blood Pressure in Patients With Primary Hypertension: a Factorial Randomized Controlled Trial.
Brief Title: Efficacy of Chlorthalidone and Hydrochlorothiazide Combined With Amiloride on Blood Pressure in Primary Hypertension.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-0553
Record Dates: First submitted 2019-04-22; First posted 2019-04-25 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Hypertension
Keywords: Hypertension; Treatment; Chlorthalidone; Hydrochlorothiazide; Amiloride
MeSH Terms: conditions — Hypertension | interventions — Chlorthalidone; Hydrochlorothiazide; Amiloride

STUDY DESIGN:
Intervention Model Description: The trial has a factorial design, where participants will receive two simultaneous interventions: a thiazide diuretic (chlorthalidone 25 mg or hydrochlorothiazide 50 mg) and a potassium-sparing diuretic (amiloride 10 mg or amiloride 20 mg). Randomization will be done in 1:1:1:1 ratio, and participants will be randomly assigned to four groups: a) chlorthalidone 25 mg + amiloride 10 mg; b) chlorthalidone 25 mg + amiloride 20 mg; c) hydrochlorothiazide 50 mg + amiloride 10 mg; and d) hydrochlorothiazide 50 mg + amiloride 20 mg.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study medication will have the same color, taste, consistency, odor and appearance. In this way, patients, care providers, outcome assessors and the entire research team will be blinded regarding the allocation to the treatment groups throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Chlorthalidone 25 mg + amiloride 20 mg (Experimental): Chlorthalidone 25 mg plus amiloride 20 mg combined in a single capsule, taken orally in the morning, for 12 weeks.
  Interventions: Drug: Chlorthalidone 25 mg; Drug: Amiloride 20 mg
- Chlorthalidone 25 mg + amiloride 10 mg (Active Comparator): Chlorthalidone 25 mg plus amiloride 10 mg combined in a single capsule, taken orally in the morning, for 12 weeks.
  Interventions: Drug: Chlorthalidone 25 mg; Drug: Amiloride 10 mg
- Hydrochlorothiazide 50 mg + amiloride 20 mg (Active Comparator): Hydrochlorothiazide 50 mg plus amiloride 20 mg combined in a single capsule, taken orally in the morning, for 12 weeks.
  Interventions: Drug: Hydrochlorothiazide 50 mg; Drug: Amiloride 20 mg
- Hydrochlorothiazide 50 mg + amiloride 10 mg (Active Comparator): Hydrochlorothiazide 50 mg plus amiloride 10 mg combined in a single capsule, taken orally in the morning, for 12 weeks.
  Interventions: Drug: Hydrochlorothiazide 50 mg; Drug: Amiloride 10 mg

INTERVENTIONS:
Drug: Chlorthalidone 25 mg — Chlorthalidone 25 mg taken orally in the morning for 12 weeks.
  Other Names: Chlorthalidone
  Arms: Chlorthalidone 25 mg + amiloride 10 mg; Chlorthalidone 25 mg + amiloride 20 mg
Drug: Hydrochlorothiazide 50 mg — Hydrochlorothiazide 50 mg taken orally in the morning for 12 weeks.
  Other Names: Hydrochlorothiazide
  Arms: Hydrochlorothiazide 50 mg + amiloride 10 mg; Hydrochlorothiazide 50 mg + amiloride 20 mg
Drug: Amiloride 20 mg — Amiloride 20 mg taken orally in the morning for 12 weeks.
  Other Names: Amiloride
  Arms: Chlorthalidone 25 mg + amiloride 20 mg; Hydrochlorothiazide 50 mg + amiloride 20 mg
Drug: Amiloride 10 mg — Amiloride 10 mg taken orally in the morning for 12 weeks.
  Other Names: Amiloride
  Arms: Chlorthalidone 25 mg + amiloride 10 mg; Hydrochlorothiazide 50 mg + amiloride 10 mg

SUMMARY:
Thiazide diuretics have demonstrated favorable blood pressure lowering efficacy, safety profile and low cost, but it is still unclear what are the equivalence of doses of their more common agents, chlorthalidone and hydrochlorothiazide. Besides, concernments about adverse metabolic effects such as hypokalemia, hyperglycemia and hyperlipidemia do exist, which may be attenuated with the concomitant administration of a potassium-sparing diuretic, such as amiloride. In addition to control adverse effects of thiazides, amiloride could offer an additional blood pressure lowering effect, but the efficacy of different doses was not fully established. This study aims to investigate the blood pressure lowering efficacy of chlorthalidone and hydrochlorothiazide, in combination with amiloride in different doses, for the initial management in patients with primary hypertension.

DETAILED DESCRIPTION:
This is a factorial (2x2) randomized double-blinded clinical trial comparing the association of a thiazide diuretic (chlorthalidone 25 mg/day or hydrochlorothiazide 50 mg/day) with a potassium-sparing diuretic (amiloride 10 mg/day or amiloride 20 mg/day) as first drug option in patients aged 30 to 75 years with primary hypertension. The thiazide diuretic and amiloride will be combined in a single capsule. The capsules will be of the same size and color, so that neither the researcher nor the patients can distinguish the treatment by their appearance. The primary outcome will be the mean change from baseline in 24-h systolic and diastolic blood pressure measured by ambulatory blood pressure monitoring (ABPM). The secondary outcomes will be the mean change from baseline in daytime and nighttime systolic and diastolic blood pressure measured by ABPM, mean change from baseline in systolic and diastolic blood pressure measured by office blood pressure, incidence of adverse events, variation of laboratory parameters and proportion of patients who achieved blood pressure control (<140/90 mmHg and <130/80 mmHg for office blood pressure and 24-h ABPM, respectively). The follow-up will last 12 weeks. For a P alpha of 0.05, power of 80%, and standard deviation of 9 mmHg, and absolute difference of 6 mmHg on systolic blood pressure on 24-h ABPM, it will be necessary to study a total of 76 patients. The sample size will be increased by 10% to compensate losses, resulting in 84 patients being randomized in total (42 for each arm).

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 30 to 75 years).
* Diagnosis of primary hypertension based on ABPM (mean 24-h systolic BP ≥130 mmHg or mean 24-h diastolic BP ≥80 mmHg).
* No current use of antihypertensive medication.

Exclusion Criteria:

* Low life expectancy.
* Other indications for the use of diuretics.
* Intolerance or contraindications to the study drugs.
* Cardiovascular disease (heart failure, myocardial infarction or stroke).
* Secondary hypertension.
* Chronic kidney disease and / or abnormal renal function (creatinine >1.5 mg/dL).
* Hyperkalemia (serum potassium >5.5 mEq/L).
* Gout.
* Previous antihypertensive treatment with more than one drug.
* Systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg measured through office blood pressure.
* Pregnancy or prospective pregnancy during the study.
* Lactating women.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2019-11-13 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in 24-h systolic blood pressure measured by ABPM. | 12 weeks
  Difference between the treatment arms in mean change from baseline in 24-h systolic blood pressure measured by ABPM.
Mean change from baseline in 24-h diastolic blood pressure measured by ABPM. | 12 weeks
  Difference between the treatment arms in mean change from baseline in 24-h diastolic blood pressure measured by ABPM.

SECONDARY OUTCOMES:
Mean change from baseline in daytime and nighttime blood pressure measured by ABPM. | 12 weeks
  Difference between the treatment arms in mean change from baseline in daytime and nighttime systolic and diastolic blood pressure measured by ABPM.
Mean change from baseline in systolic and diastolic blood pressure measured by office blood pressure. | 12 weeks
  Difference between the treatment arms in mean change from baseline in systolic and diastolic blood pressure measured by office blood pressure.
Proportion of participants reporting adverse events. | 12 weeks
  Difference between treatment arms in the proportion of participants reporting adverse events.
Mean change from baseline in total cholesterol. | 12 weeks
  Difference between the treatment arms in mean change from baseline in serum total cholesterol, measured in mg/dL.
Mean change from baseline in HDL cholesterol (HDL-C). | 12 weeks
  Difference between the treatment arms in mean change from baseline in serum HDL cholesterol (HDL-C), measured in mg/dL.
Mean change from baseline in LDL cholesterol (LDL-C). | 12 weeks
  Difference between the treatment arms in mean change from baseline in serum LDL cholesterol (LDL-C), measured in mg/dL.
Mean change from baseline in triglycerides. | 12 weeks
  Difference between the treatment arms in mean change from baseline in serum triglycerides, measured in mg/dL.
Mean change from baseline in creatinine. | 12 weeks
  Difference between the treatment arms in mean change from baseline in serum creatinine, measured in mg/dL.
Mean change from baseline in urea. | 12 weeks
  Difference between the treatment arms in mean change from baseline in serum urea, measured in mg/dL.
Mean change from baseline in potassium. | 12 weeks
  Difference between the treatment arms in mean change from baseline in serum potassium, measured in mEq/L.
Mean change from baseline in sodium. | 12 weeks
  Difference between the treatment arms in mean change from baseline in serum sodium, measured in mg/dL.
Mean change from baseline in magnesium. | 12 weeks
  Difference between the treatment arms in mean change from baseline in serum magnesium, measured in mg/dL.
Mean change from baseline in uric acid. | 12 weeks
  Difference between the treatment arms in mean change from baseline in serum uric acid, measured in mg/dL.
Mean change from baseline in fasting plasma glucose. | 12 weeks
  Difference between the treatment arms in mean change from baseline in fasting plasma glucose, measured in mg/dL.
Mean change from baseline in hemoglobin A1c (HbA1c). | 12 weeks
  Difference between the treatment arms in mean change from baseline in hemoglobin A1c (HbA1c), measured in percentage.
Proportion of participants achieving blood pressure control. | 12 weeks.
  Difference between treatment arms in the proportion of participants achieving blood pressure control. Blood pressure control will be defined as <140/90 mmHg and <130/80 mmHg for office BP and 24-h ABPM, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Fuchs, MD, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
This trial is in accordance with the compliance of the reproducibility standards accordingly to the International Committee of Medical Journal Editors (ICMJE). The investigators intend to publish the results in an open-access journal, indexed at the Directory of Open Access Journals, with the copyrights transferred to the authors (CC By 4.0). Also, all materials, raw and treated data, statistical code and outputs will be publicly shared without restrictions to access the data neither expiration date. The repository was not chosen yet and will be provided in further amendments or in the final report of this study. All laboratory specimens, reports, data collection, process, and administrative forms will be identified by a coded identification number to maintain participant confidentiality. After full data analysis, all subject identifiers will be erased.
Time Frame: The individual participant dataset will become available at a public repository up to six months after the first study publication.
Access Criteria: A simple registration will grant access to study datasets. The website for these files is not defined at the time of registration.

REFERENCES:
- [Derived] Martins VM, Helal L, Ferrari F, Bottino LG, Fuchs SC, Fuchs FD. Efficacy of chlorthalidone and hydrochlorothiazide in combination with amiloride in multiple doses on blood pressure in patients with primary hypertension: a protocol for a factorial randomized controlled trial. Trials. 2019 Dec 16;20(1):736. doi: 10.1186/s13063-019-3909-z. PMID 31843024